CLINICAL TRIAL: NCT03939793
Title: Combining Best Practices for Health Behavior Change: a Randomized Controlled Trial of Digital Health, Financial Incentives and Community Health Worker Support for Vulnerable Populations
Brief Title: Using Digital Health, Financial Incentives, and Community Health Worker Support to Change Health Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: The Commonwealth Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20191985
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus
Keywords: Community Health Worker; Financial Incentives
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Clinical Support (Placebo Comparator): Participants will continue with their usual diabetes care provided by their clinic. Participants will receive a free wireless glucometer on the day of enrollment if they do not already have one.
  Interventions: Other: Usual Care
- DFI Alone (Active Comparator): Participants will receive a free wireless glucometer on the day of enrollment if they don't already have one. To encourage habit formation, for the first 6 weeks of the trial, participants will be eligible for a daily lottery incentive for every day that they use their glucometer. Investigators will use an approach similar to what we have used in prior DFI trials: the lottery will provide infrequent large payoffs (a 1 in 100 chance of a US$50 reward) and more frequent small payoffs (an 18 in 100 chance of a US $5 reward). Participants who draw the winning lottery number, but did not check their glucose the day prior will receive an automated text or e-mail message informing them what earnings they would have won had they used their glucometer. After 6 weeks, investigators will terminate the lottery but continue to monitor patients' adherence to glucose self-monitoring.
  Interventions: Behavioral: Digital health monitoring with financial incentives
- Hybrid DFI CHW (Experimental): Participants in the hybrid intervention will receive a wireless glucometer if they don't already have one and financial incentives just as in the DFI intervention. However, any individuals who have low adherence (no self-monitoring) or elevated glucose readings (>300 mg/dL) for >30% of days over any 2 week period in the first 12 weeks of the study will be assigned to receive ongoing community health worker (CHW) support for the duration of the 24-week study period.
  Interventions: Behavioral: IMPaCT Community Health Worker; Behavioral: Digital health monitoring with financial incentives

INTERVENTIONS:
Behavioral: IMPaCT Community Health Worker — Once a CHW receives notification of a struggling patient, the CHW will visit the patient at their home within 1-2 days to initiate the IMPaCT intervention.
  1. Elements of the standard IMPaCT intervention: During the first home visit, the CHW will use an in-depth semi-structured interview guide to get to know patients holistically and assess for unmet socioeconomic needs. This allows patients to express goals in line with their own needs and preferences. These individualized goals will become the basis for tailored action plans. The CHW will then provide hands-on, tailored support for the remainder of the 24-week study period to help patients achieve their goals.
  2. Additional elements to help patients cope with failure: In this study, we will test a refined version of IMPaCT that incorporates two behavioral techniques for coping with failure: positive affect induction and attribution retraining.
  Arms: Hybrid DFI CHW
Behavioral: Digital health monitoring with financial incentives — Participants are encouraged to use their glucometer to check their blood glucose via bidirectional texting and lottery-based financial incentives, which both serve to reinforce self-monitoring behavior.
  Arms: DFI Alone; Hybrid DFI CHW
Other: Usual Care — Usual Care
  Arms: Usual Clinical Support

SUMMARY:
This randomized controlled trial tests how digital health monitoring with financial incentives (DFI) and community health worker (CHW) support may affect how a person manages their diabetes. Participants will be randomized to one of three arms: 1) DFI intervention, 2) hybrid DFI/CHW intervention, or 3) usual care. Investigators hypothesize that compared to usual care and DFI alone, the hybrid intervention will lead to more glucose self-monitoring and greater improvements in glycosylated hemoglobin.

DETAILED DESCRIPTION:
Low-income Americans struggle to stay healthy in the face of real-life challenges such as housing insecurity or trauma. Two interventions show promise for promoting behavior change and improving health outcomes: digital health interventions coupled with financial incentives (DFI) and community health workers (CHWs). Yet, these interventions have limitations; DFI interventions have low uptake and high attrition among vulnerable populations, while CHW interventions are relatively resource intensive.

Investigators propose a 24-week randomized trial of a hybrid DFI/CHW intervention among a population of 150 low-income patients with diabetes. Participants will be randomized to one of three arms: 1) DFI intervention, 2) hybrid DFI/CHW intervention, 3) usual care. Participants assigned to DFI will receive a free wireless glucometer and be eligible for a lottery incentive if they use their glucometer. Participants assigned to the hybrid DFI/CHW intervention will receive the same glucometer and incentives. If they exhibit low adherence to self-monitoring or poor glucose control, they will also receive support from a CHW who would help patients to address underlying socioeconomic barriers and cope with setbacks. Investigators hypothesize that compared to usual care and DFI alone, the hybrid intervention will lead to more glucose self-monitoring and greater improvements in glycosylated hemoglobin.

ELIGIBILITY:
Inclusion Criteria:

* Penn Medicine patients diagnosed with diabetes mellitus.
* Glycosylated hemoglobin >=9% within the past 6 months.
* Requires insulin.
* Uninsured/publicly insured.
* Residents of high-poverty ZIP codes in West/Southwest Philadelphia.
* Have access to a cellphone with unlimited text message capabilities.

Exclusion Criteria:

* Already have a continuous glucose monitor.
* Previously enrolled in the study.
* Currently have an outpatient CHW.
* Unwilling/unable to provide informed consent.
* In another study that asks participants to monitor their blood sugar.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitehouse CR, Knowles M, Long JA, Mitra N, Volpp KG, Xu C, Sabini C, Gerald N, Estrada I, Jones D, Kangovi S. Digital Health and Community Health Worker Support for Diabetes Management: a Randomized Controlled Trial. J Gen Intern Med. 2023 Jan;38(1):131-137. doi: 10.1007/s11606-022-07639-6. Epub 2022 May 17. PMID 35581452

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Participants randomized to the usual-care arm were asked to check their daily blood glucose and to continue with their usual care.
- Digital Health: Participants randomized to the digital health arm were asked to check their blood glucose and text the value daily to a phone number linked to the Way to Health platform. To promote early motivation and habit formation, participants were entered into a lottery each day they texted their glucose values for the first 6 weeks of the study period. Each day participants texted, the lottery provided an 18 in 100 chance of winning $5 and 1 in 100 chance of winning $50. Accrued money was distributed to participants biweekly on a reloadable card.
  If participants texted in a blood glucose value that was pre-established as medically dangerous (< 60, > 400), they received an automated text encouraging them to follow up with their provider. These values were also routed directly to the study clinician who called each patient within 24 hours to provide clinical management and coordinate care with the patient's provider.
- Hybrid Digital Health and Community Health Worker Support: Participants in the hybrid arm received all aspects of the digital health intervention. Additionally, CHWs met with participants at enrollment and provided brief coaching using positive affect induction and attribution retraining to increase resilience to setbacks. At this meeting, CHWs explained to patients that they might work with them in the future if they needed additional support. During the first 12 weeks of the study, hybrid arm participants with low rates of SMBG (defined as 5 instances of missed readings) and/or elevated glucose readings (defined as a glucose level > 300 mg/dL for > 30% of days over any 2-week period) were 'escalated' to receive intensive CHW support.
  CHWs implemented the IMPaCT intervention, in which the CHW used an in-depth semi-structured interview guide to get to know participants' strengths, goals, and unmet social needs. Participants' individualized goals became the basis for tailored action plans. For the remainder of the 24-week study period, CHWs provided coaching, social support, advocacy, and navigation to support participants in achieving their health goals. CHWs communicated with participants at least once per week, including monthly face-to-face contact. CHWs normalized setbacks and used positive affect induction and attribution retraining to help patients to cope with failure. CHWs also helped participants connect to long-term family and social supports after the intervention ended.
Period: Overall Study
Arm/Group | Usual Care | Digital Health | Hybrid Digital Health and Community Health Worker Support
Started | 50 | 50 | 50
Completed | 40 | 34 | 28
Not Completed | 10 | 16 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Digital Health | Hybrid Digital Health and Community Health Worker Support | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (8.7) | 55.0 (14.1) | 54.1 (12.8) | 55.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participant declined to answer
  Participants
    number analyzed (Participants) | 49 | 50 | 50 | 149
    Female | 34 | 36 | 35 | 105
    Male | 15 | 14 | 15 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 8
  Not Hispanic or Latino | 48 | 46 | 47 | 141
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 4 | 5
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 45 | 39 | 42 | 126
  White | 1 | 0 | 3 | 4
  More than one race | 2 | 3 | 0 | 5
  Unknown or Not Reported | 2 | 6 | 1 | 9
Highest level of education [Count of Participants; unit: Participants]
  Less than HS | 15 | 10 | 11 | 36
  HS or GED | 16 | 22 | 20 | 58
  Some college/technical school | 15 | 13 | 14 | 42
  College graduate | 4 | 5 | 5 | 14
Household income [Count of Participants; unit: Participants]
  <15K | 32 | 30 | 32 | 94
  >=15K | 16 | 18 | 17 | 51
  Unknown | 2 | 2 | 1 | 5
Employed [Count of Participants; unit: Participants] | 9 | 7 | 2 | 18
Insurance [Count of Participants; unit: Participants]
  Medicaid | 27 | 27 | 33 | 87
  Medicaid/Medicare | 23 | 22 | 16 | 61
  Uninsured | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 1
Prior healthcare utilization, past 6 months (self-report) [Count of Participants; unit: Participants]
  Any ED visit | 23 | 29 | 30 | 82
  Any hospital admission | 19 | 20 | 14 | 53
Postponed needed medical care [Count of Participants; unit: Participants] — Response to question: "Was there any time during the past 12 months when you put off or postponed getting medical care you thought you needed?"
  Participants | 7 | 9 | 11 | 27
Health literacy [Mean (Standard Deviation); unit: units on a scale] — Single Item Literacy Screener (SILS): "How often do you need to have someone help you when you read instructions, pamphlets, or other written material from your doctor or pharmacy?", response options Never, Rarely, Sometimes, Often, Always. Score range: 1-5, with higher scores indicating lower health literacy.
  units on a scale | 1.9 (1.1) | 1.8 (1.2) | 2.1 (1.3) | 1.9 (1.2)
More than 1 competing need [Count of Participants; unit: Participants] — Basic needs scale measuring difficulty accessing the following needs: shelter, food, washing, bathroom, transportation, and telephone. Reported needs summed to generate score; score of 2 or more indicates more than one competing need.
  Participants | 14 | 23 | 20 | 57
Drug use [Count of Participants; unit: Participants] | 8 | 6 | 5 | 19
Alcohol overuse [Count of Participants; unit: Participants] | 11 | 10 | 7 | 28
Adverse childhood experiences [Mean (Standard Deviation); unit: units on a scale] — Experiences include 10 forms of abuse (physical, emotional, sexual), neglect (physical, emotional), and household instability (household member with mental illness, household member with substance use disorder, household member incarcerated, domestic violence, loss of a parent). Number of reported experiences summed to generate a score of 0-10 with highest score indicating most experiences.
  units on a scale | 3.1 (2.8) | 3.3 (2.6) | 2.8 (2.4) | 3.0 (2.6)
Perceived stress [Mean (Standard Deviation); unit: units on a scale] — Perceived stress scale (PSS-4) assesses respondent's perceptions of stress over the last month, including feelings of lack of control, ability to handle personal problems, things going their way, and difficulties unable to be overcome. Score range: 0-16, with the highest score indicating high stress.
  units on a scale | 5.9 (3.5) | 6.1 (4.0) | 5.7 (3.6) | 5.9 (3.7)
Low social support [Count of Participants; unit: Participants] — ENRICHD Social Support Instrument (ESSI) measures respondent's range of social support, including someone available to listen to problems, give advice, support with chores, etc.; total scores range from 8 to 34; higher scores equal higher levels of support. Low social support defined as total score of 18 or less and scoring 2 or less on at least 2 items.
  Participants | 4 | 7 | 7 | 18
HbA1C [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] | 10.94 (2.21) | 11.05 (1.58) | 10.89 (2.01) | 10.96 (1.94)
Patient Activation Measure [Mean (Standard Deviation); unit: units on a scale] — Patient Activation Measure - 13 assesses patient knowledge, skill, and confidence for self-management of health conditions. Scored from 0-100; higher scores indicated higher levels of knowledge, skill, and confidence for health self-management.
  units on a scale | 69.5 (16.6) | 67.3 (15.4) | 65.8 (14.2) | 67.6 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Glucose Self-monitoring Adherence
Description: constructed by summing the number of days in the study period that the glucometer was used divided by the total number of days in study period
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Usual Care | Digital Health | Hybrid Digital Health and Community Health Worker Support
Number analyzed (Participants) | 40 | 34 | 28
percentage of days | 65 (28) | 70 (25) | 72 (29)

2. Other Pre Specified Outcome: Change in Glycosylated Hemoglobin
Description: Change in glycosylated hemoglobin from baseline to 6 month follow-up assessment.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Usual Care | Digital Health | Hybrid Digital Health and Community Health Worker Support
Number analyzed (Participants) | 23 | 21 | 24
percentage of glycosylated hemoglobin | -0.49 (1.75) | -0.85 (1.90) | -0.74 (1.66)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 6 months post-enrollment.
Arm/Group | Usual Care | Digital Health | Hybrid Digital Health and Community Health Worker Support
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 13/50 | 13/50 | 14/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=50) | Digital Health (N=50) | Hybrid Digital Health and Community Health Worker Support (N=50)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1 | 0
Volume Overload (Cardiac disorders) | 1 | 0 | 0
Diabetic Ketoacidosis (Endocrine disorders) | 0 | 0 | 1
Hyperglycemia (Endocrine disorders) | 2 | 1 | 1
Hypoglycemia (Endocrine disorders) | 0 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 1 | 1
Altered mental status (Nervous system disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Finger infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0
Post-operative pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Seizure (Nervous system disorders) | 2 | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1 | 0
Intrauterine fetal demise (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Pyelonephritis (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure with hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Stroke (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The COVID pandemic may have led to a higher-than-expected rate of loss to follow-up at 6 months. A COVID-19 modification truncated our primary outcome from 6 to 3 months. Unlike many DHI requiring smartphones, we only required participants to have a basic cell phone; participants needed to text their SMBG to the study platform which may have increased attrition. Because we used low-tech glucometers covered by Medicaid, we extracted data from the physical device, resulting in some missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT03939793/Prot_SAP_000.pdf